CLINICAL TRIAL: NCT02497469
Title: A Randomized, Double-Blind, Double-Dummy, Multicenter, Active-Controlled Study to Evaluate the Efficacy and Safety of Vedolizumab IV Compared to Adalimumab SC in Subjects With Ulcerative Colitis
Brief Title: An Efficacy and Safety Study of Vedolizumab Intravenous (IV) Compared to Adalimumab Subcutaneous (SC) in Participants With Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MLN0002-3026; U1111-1168-6713 (Registry Identifier: WHO); 2015-000939-33 (EudraCT Number); NL54690.056.15 (Registry Identifier: CCMO)
Record Dates: First submitted 2015-07-10; First posted 2015-07-14 (Estimated); Results first posted 2019-10-10 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Colitis, Ulcerative
Keywords: Drug Therapy
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vedolizumab IV 300 mg (Experimental): Vedolizumab 300 milligram (mg), infusion, intravenously over 30 minutes on Day 1 and Weeks 2, 6, 14, 22, 30, 38, and 46. Adalimumab placebo-matching injection, subcutaneously on Day 1, Week 2, and every 2 weeks thereafter up to Week 50.
  Interventions: Drug: Vedolizumab; Drug: Adalimumab placebo
- Adalimumab SC 160/80/40 mg (Active Comparator): Adalimumab 160 mg, injection, subcutaneously on Day 1, adalimumab 80 mg, injection, subcutaneously at Week 2, then adalimumab 40 mg, injection, subcutaneously every 2 weeks thereafter up to Week 50. Vedolizumab placebo-matching infusion, intravenously on Day 1 and Weeks 2, 6, 14, 22, 30, 38, and 46.
  Interventions: Drug: Adalimumab; Drug: Vedolizumab placebo

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab infusion
  Arms: Vedolizumab IV 300 mg
Drug: Adalimumab placebo — Adalimumab placebo-matching injection
  Arms: Vedolizumab IV 300 mg
Drug: Adalimumab — Adalimumab injection
  Arms: Adalimumab SC 160/80/40 mg
Drug: Vedolizumab placebo — Vedolizumab placebo-matching infusion
  Arms: Adalimumab SC 160/80/40 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of vedolizumab intravenous (IV) treatment compared to adalimumab subcutaneous (SC) treatment over a 52-week treatment period.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. Vedolizumab is being tested to treat people who have ulcerative colitis. This study will look at the stool frequency, rectal bleeding and findings on endoscopy of people who take vedolizumab compared to those who take adalimumab.

The study will enroll approximately 658 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Vedolizumab 300 mg IV
* Adalimumab 160 mg on Day 1 followed by 80 mg on Week 2 then 40 mg every 2 weeks SC

All participants will receive 1 intravenous infusion on Day 1 and Weeks 2, 6, 14, 22, 30, 38, and 46. All participants will also receive 4 SC injections on Day 1 or 2 SC injections each on Days 1 and 2, followed by 2 SC injections in 1 day on Week 2 and then 1 SC injection every 2 weeks for up to Week 50. All participants will be asked to record the symptoms of ulcerative colitis in a daily diary.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is 79 weeks. Participants will make approximately 11 visits to the clinic, and will be contacted by telephone 6 months after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of ulcerative colitis established at least 3 months prior to screening by clinical and endoscopic evidence and corroborated by a histopathology report.
2. Has moderately to severely active ulcerative colitis as determined by a Mayo score of 6 to 12 with an endoscopic subscore greater than or equal to >=2 within 14 days prior to the randomization.
3. Has evidence of ulcerative colitis proximal to the rectum (>=15 centimeter [cm] of involved colon).
4. With extensive colitis (up to the hepatic flexure) or pancolitis of >8 years duration or left-sided colitis of >12 years duration must have documented evidence that a surveillance colonoscopy was performed within 12 months of the initial screening visit (may be performed during the Screening Period).
5. The participant:

   1. Has had previous treatment with tumor necrosis factor- alpha (TNF-alpha) antagonists without documented clinical response to treatment (example, due to lack of response [primary nonresponders], loss of response, or intolerance [secondary nonresponders]), or
   2. Has previously used a TNF-alpha antagonists (except adalimumab), and discontinued its use due to reasons other than safety, or
   3. Is naïve to TNF-alpha antagonist therapy but is failing current treatment (example, corticosteroids, 5-aminosalicylate [5-ASA], or immunomodulators).

Exclusion Criteria:

1. Clinical evidence of abdominal abscess or toxic megacolon at Screening.
2. Has had an extensive colonic resection, subtotal or total colectomy.
3. Has had ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine.
4. Has a diagnosis of Crohn's colitis or indeterminate colitis, ischemic colitis, radiation colitis, diverticular disease associated with colitis, or microscopic colitis.
5. Has received any of the following for the treatment of underlying disease within 30 days of randomization:

   1. Non-biologic therapies (example, cyclosporine, tacrolimus, thalidomide) other than those specifically listed in Section Permitted Medications For Treatment of UC.
   2. An approved non-biologic therapy in an investigational protocol.
6. Has received any investigational or approved biologic or biosimilar agent within 60 days or 5 half lives prior to the screening (whichever is longer).
7. Has previously received natalizumab, efalizumab, adalimumab, AMG-181, anti-mucosal addressin cell adhesion molecule-1 antibodies, or rituximab.
8. Has previously received vedolizumab.
9. Has history or evidence of adenomatous colonic polyps that have not been removed, or colonic mucosal dysplasia.
10. Evidence of an active infection during Screening.
11. Evidence of, or treatment for, Clostridium difficile (C. difficile) or other intestinal pathogen within 28 days prior to the 1st dose of study drug.
12. Has chronic hepatitis B virus (HBV) infection* or chronic hepatitis C virus (HCV) infection (* HBV immune participants, ie, being hepatitis B surface antigen [HBsAg], may participate).
13. Has active or latent TB, regardless of treatment history.
14. Has used a topical (rectal) treatment with (5-ASA) or corticosteroid enemas/suppositories within 2 weeks of the administration of the 1st dose of study drug.
15. Has a positive progressive multifocal leukoencephalopathy (PML) subjective symptom checklist prior to the administration of the first dose of study drug.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 771 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2019-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (329):
- United States (77):
  - IMC - Diagnostic and Medical Clinic, Mobile, Alabama
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - Arkansas Primary Care Clinic, PA, Little Rock, Arkansas
  - WCCT Global (PH 1 Unit), Costa Mesa, California
  - California Medical Research Associates Inc., Northridge, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Rocky Mountain Gastroenterology, Lakewood, Colorado
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Innovative Medical Research of South Florida, Inc., Aventura, Florida
  - Advanced Clinical Research of Miami, Doral, Florida
  - Wellness Clinical Research, Hialeah Gardens, Florida
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - Gastro Health, Miami, Florida
  - Medical Professional Clinical Research, Miami, Florida
  - Tellus Clinical Research, Inc., Miami, Florida
  - South Florida Research Phase I-IV, Miami Springs, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - BRCR Medical Center, Inc., Plantation, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Gastroenterology of Southern Associates, New Albany, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - University of Louisville, Louisville, Kentucky
  - Research Concierge, LLC, Owensboro, Kentucky
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Lafayette General Medical Center, Lafayette, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Digestive Disease Associates, Catonsville, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Center for Digestive Health and Nutritional Excellence, Troy, Michigan
  - Gastroenterology Associates of Western Michigan, P.L.C., Wyoming, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Digestive Health Center PA, Ocean Springs, Mississippi
  - Ehrhardt Clinical Research, LLC, Belton, Missouri
  - Truman Medical Centers, Inc., Kansas City, Missouri
  - Alegent Creighton Clinic Gastroenterology, Omaha, Nebraska
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - Long Island Clinical Research Associates, Great Neck, New York
  - Mount Sinai - PRIME, Lake Success, New York
  - Digestive Disease Care, New Hyde Park, New York
  - Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Consultants for Clinical Research Inc., Cincinnati, Ohio
  - Ohio State University Clinical Trials Management Office, Columbus, Ohio
  - Dayton Gastroenterology, Inc, Dayton, Ohio
  - Gastro-Enterology Research of Lima, Lima, Ohio
  - Options Health Research, Tulsa, Oklahoma
  - The Oregon Clinic-West Hills Gastroenterology, Portland, Oregon
  - Main Line Gastroenterology Associates, Malvern, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Invocare Clinical Research Center, West Columbia, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Digestive Disease Consultants - Dallas, Dallas, Texas
  - Baylor University Hospital, Dallas, Texas
  - MedResearch, Inc, El Paso, Texas
  - Gastroenterology Consultants of South Texas, PA, Harlingen, Texas
  - Gulf Coast Research Group LLC, Houston, Texas
  - Texas Digestive Disease Consultants - Irving, Irving, Texas
  - Advanced Clinical Research Associates, Plano, Texas
  - Gastroenterology Research of San Antonio, LLC, San Antonio, Texas
  - Texas Digestive Disease Consultants - Southlake, Southlake, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Virginia Mason Seattle Main Clinic, Seattle, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Allegiance Research Specialists, LLC, Milwaukee, Wisconsin
- Argentina (4):
  - Instituto de Investigaciones Clinicas-Mar del Plata, Mar del Plata, Buenos Aires
  - Instituto Medico CER, Quilmes, Buenos Aires
  - Expertia S.A- Mautalen Salud e Investigacion, Ciudad Autonoma Buenos Aires
  - Centro de Investigaciones Clinicas Instituto del Corazon, Córdoba
- Australia (8):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Mater Adult Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Tennyson Centre Day Hospital, Bedford Park, South Australia
  - Ballarat Base Hospital, Ballarat, Victoria
  - Monash Medical Centre Moorabbin, Clayton, Victoria
  - St Frances Xavier Cabrini Hospital, Malvern, Victoria
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Bosnia and Herzegovina (3):
  - University Clinical Centre of the Republic of Srpska, Banja Luka
  - University Clinical Hospital Mostar, Mostar
  - University Clinic Centre Sarajevo, Sarajevo
- Bulgaria (13):
  - MHAT - Pazardzhik AD, Pazardzhik
  - MHAT 'Avis Medica' OOD, Pleven
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - MHAT "Hadzhi Dimitar", OOD, Sliven
  - "City Clinic UMHAC" EOOD, Sofia
  - Medical Center "Excelsior", OOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - UMHAT 'Tsaritsa Yoanna - ISUL', EAD, Sofia
  - Fourth MHAT - Sofia EAD, Sofia
  - Military Medical Academy - MHAT - Sofia, Sofia
  - UMHAT 'Sveta Anna' AD, Sofia
  - Medical Center "Nov Rehabilitatsionen Tsentar", EOOD, Stara Zagora
  - MHAT 'Sv. Marina', EAD, Varna
- Canada (7):
  - University of Alberta, Edmonton, Alberta
  - McMaster University Health Sciences Center, Hamilton, Ontario
  - Hotel Dieu Hospital, Kingston, Ontario
  - LHSC - University Hospital, London, Ontario
  - LHSC - Victoria Hospital, London, Ontario
  - Toronto Digestive Disease Associates, Inc., Vaughan, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan
- Colombia (2):
  - Fundacion Oftalmologica de Santander - FOSCAL, Floridablanca
  - Instituto de Coloproctologia ICO S.A.S., Medellín
- Croatia (7):
  - Clinical Hospital Centre Osijek, Osijek
  - General Hospital Pula, Pula
  - Polyclinic Medico, Rijeka
  - Clinical Hospital Center "Sestre Milosrdnice", Zagreb
  - Clinical Hospital Centre Zagreb, Zagreb
  - Clinical Hospital Dubrava, Zagreb
  - Clinical Hospital Merkur, Zagreb
- Czechia (9):
  - CCBR - Brno - CZ, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - CCBR Czech, a.s, Pardubice
  - A-Shine, Pilsen
  - CCBR - Prague - CZ, Prague
  - Klinicke centrum ISCARE Lighthouse, Prague
  - Axon Clinical, s.r.o., Prague
  - Thomayerova nemocnice, Praha 4 - Krc
- Denmark (4):
  - Nordsjallands Hospital, Frederikssund, Frederikssund
  - Hvidovre_Hospital, Hvidovre
  - Koge Sygehus, Køge
  - Odense Universitetshospital, Odense C
- Estonia (3):
  - West Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- France (11):
  - CHU Nice - Hopital de l'Archet 2, Nice, Alpes Maritimes
  - Hopital Saint Joseph, Marseille, Bouches-du-Rhone
  - Hopital Nord - CHU Marseille, Marseille, Bouches-du-Rhone
  - Groupe Hospitalier Sud - Hopital Haut-Leveque, Pessac, Gironde
  - CHU de Toulouse - Hopital Rangueil, Toulouse, Haute Garonne
  - Hopital Beaujon, Clichy, Hauts De Seine
  - Hopital de Brabois Adultes, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - Hopital Claude Huriez - CHU Lille, Lille, Nord
  - CHU Saint Etienne - Hopital Nord, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - CHU Amiens - Hopital Sud, Amiens, Somme
  - Centre Hospitalier Departemental Les Oudairies, La Roche S/ Yon Cedex 9, Vendee
- Germany (12):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main, Hesse
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz, Rhineland-Palatinate
  - EUGASTRO GmbH, Leipzig, Saxony
  - Universitaetsklinikum Magdeburg A.oe.R, Magdeburg, Saxony-Anhalt
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck, Schleswig-Holstein
  - Charite - Campus Virchow-Klinikum, Berlin
  - Krankenhaus Waldfriede e. V., Berlin
  - Asklepios Klinik Hamburg, Hamburg
- Hong Kong (3):
  - The University of Hong Kong, Hong Kong
  - Tuen Mun Hospital, Medicine & Geriatrics
  - The Chinese University of Hong Kong, Shatin
- Hungary (9):
  - Bekes Megyei Kozponti Korhaz Dr. Rethy Pal Tagkorhaza, Békéscsaba
  - Peterfy Sandor utcai Korhaz-Rendelointezet es Baleseti Kozpont, Budapest
  - Semmelweis Egyetem, Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger
  - Pecsi Tudomanyegyetem, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
- Israel (11):
  - HaEmek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Hillel Yaffe Medical, Hadera
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Clalit Health Services-Lev Talpiyot, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Center, Nahariya
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (16):
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Istituto Clinico Humanitas, Rozzano, Milano
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese, Milano
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Ospedaliera Ospedale Cannizzaro, Catania
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli (Presidio Ospedale Sacco), Milan
  - A.O.U. Policlinico di Modena, Modena
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Seconda Universita degli Studi di Napoli, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliera Vincenzo Cervello, Palermo
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera San Camillo Forlanini, Roma
- Latvia (2):
  - Digestive Diseases Center "Gastro", Riga
  - Pauls Stradins Clinical University Hospital SLLC, Riga
- Lithuania (4):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Klaipeda Republican Hospital, Public Institution, Klaipėda
  - Klaipeda University Hospital, Public Institution, Klaipėda
  - Vilnius University Hospital Santariskiu Clinic, Public Institution, Vilnius
- Mexico (5):
  - Morales Vargas Centro de Investigacion, S.C., León, Guanajuato
  - Centro de Investigacion Farmacologica del Bajio, S.C., León, Guanajuato
  - Christus Muguerza Sur S.A. de C.V., Monterrey, Nuevo León
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Sociedad de Metabolismo y Corazon S.C, Veracruz
- Netherlands (5):
  - Onze Lieve Vrouwe Gasthuis, Locatie Oost, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen (UMCG), Groningen
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
- Poland (17):
  - SP ZOZ Wojewodzki Szpital Zespolony im. J. Sniadeckiego, Bialystok
  - NZOZ Vitamed, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - SP CSK im. prof. K. Gibinskiego SUM, Katowice
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - SPZOZ Uniwersytecki Szpital Klin. nr 1 im.N.Barlickiego UM, Lodz
  - Santa Familia Centrum Badan, Profilaktyki i Leczenia, Lodz
  - GASTROMED Sp. z o.o., Lublin
  - SOLUMED Centrum Medyczne, Poznan
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Centrum Zdrowia Matki, Dziecka i Mlodziezy, Warsaw
  - Centralny Szpital Kliniczny MSW w Warszawie, Warsaw
  - Centrum Onkologii-Instytut im. M. Sklodowskiej Curie, Warsaw
  - Nzoz Vivamed, Warsaw
  - LexMedica Osrodek Badan Klinicznych, Wroclaw
  - Ars-Medica S.C Rybak Maria, Rybak Zbigniew, Wroclaw
  - EuroMediCare Szpital Specjalistyczny z Przychodni we Wroclawiu, Wroclaw
- Portugal (6):
  - Hospital de Braga, Braga
  - Centro Hospitalar e Universitario de Coimbra E.P.E, Coimbra
  - Centro Hospitalar Cova da Beira, Covilha
  - Hospital da Senhora da Oliveira Guimaraes, Guimarães
  - Centro Hospitalar do Alto Minho - Unidade Local de Saude do Alto Minho, EPE, Viana do Castelo
  - Centro Hospitalar Vila Nova de Gaia/Espinho, E.P.E, Vila Nova de Gaia
- Romania (3):
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - S.C Centrul de Gastroenterologie Dr. Goldis S.R.L, Timișoara
- Russia (20):
  - SBEI HPE "Kazan State Medical University" of the MoH of the RF, Kazan'
  - TSBIH "Territorial Clinical Hospital", Krasnoyarsk
  - Research Institute of Gastroenterology, Moscow
  - FSBIH "Central Clinical Hospital of Russian Academy of Sciences", Moscow
  - FSBI State Scientific Centre of Coloproctology" of the MoH of RF, Moscow
  - SBIH of Nizhniy Novgorod region " Nizhniy Novgorod Regional Clinical Hospital n.a. N.A. Semashko", Nizhny Novgorod
  - SBEIHPE Novosibirsk State Medical University, Novosibirsk
  - FSBI "Scientific Research Institute of Physyology and Basic Medicine" under the SB of RAMS, Novosibirsk
  - BHI of Omsk region Clinical Oncology Dispensary, Omsk
  - SBEI of HPE "Omsk SMA" SBEI HPE "Omsk State Medical University" of the MoH of the RF, Omsk
  - SBEI HPE "Rostov State Medical University" of the MoH of the RF, Rostov-on-Don
  - FSMEI HPE Military Medical Academy n.a. S.M.Kirov"of Ministry of Defense of Russia, Saint Petersburg
  - SPb SBIH "City Hospital of Saint Martyr Elizaveta", Saint Petersburg
  - SPb SBIH "City Hospital # 26", Saint Petersburg
  - SPb SBIH "City Hospital # 9", Saint Petersburg
  - Private Educational Institution of Higher Education "Medical University "REAVIZ", Samara
  - SIH "Regional Clinical Hospital ", Saratov
  - SPb SBIH "City Hospital # 40 of Kurortnyi region", Sestroretsk
  - RSBIH "Smolensk Regional Clinical Hospital", Smolensk
  - SBIH of Yaroslavl region " Regional Clinical Hospital ", Yaroslavl
- Serbia (7):
  - Clinical Center of Serbia, Belgrade
  - Clinical Center Zvezdara, Belgrade
  - Clinical Center Bezanijska kosa, Belgrade
  - Clinical Center Zemun, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
  - Clinical Center of Vojvodina, Novi Sad
- Slovakia (6):
  - IBDcentrum s.r.o., Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica Ruzinov, Bratislava
  - Gastroped s.r.o., Košice
  - KM Management spol. s r.o., Nitra
  - Gastro I, s.r.o., Prešov
  - Frantisek Horvath- GEA, Šahy
- South Korea (14):
  - Hanyang Univerisy Guri Hospital, Guri-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Kyungpook National University Hospital, Daegu, Gyeongsangbuk-do
  - Pusan National University Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Marys Hospital, Seoul
- Spain (4):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Ramon y Cajal, Madrid
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
- Turkey (Türkiye) (6):
  - Ankara University Medical Faculty, Ankara
  - Acibadem Fulya Hospital, Istanbul
  - Haydarpasa Numune Training and Research Hospital, Istanbul
  - Marmara University Pendik Research and Training Hospital, Istanbul
  - Kocaeli Derince Training and Research Hospital, Kocaeli
  - Mersin University Medical Faculty, Mersin
- Ukraine (20):
  - RCI Chernivtsi RCH Dep of Surgery Bukovinian SMU, Chernivtsi
  - SI Institute of Gastroenterology of NAMSU Dept of Stomach & Duodenum Diseases, D&ThN SI DMA of MoHU, Dnipropetrovsk
  - Regional CH Dep of Gastroenterology SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - CI of PH Kharkiv CCH #2, Kharkiv
  - CI A.and O. Tropiny City Clinical Hospital, Kherson
  - Treatment-Diagnostic Center of Private Enterprise of PPC Atsynus, Kirovohrad
  - CI of Kyiv RC Kyiv Regional Clinical Hospital, Kyiv
  - MI of Healthcare Kyiv RCH P.L. Shupyk NMA of PGE, Kyiv
  - Kyiv CCH #12 Dept of Therapy O.O.Bogomolets NMU, Kyiv
  - Kyiv CCH #8 Dept of Gastroenterology P.L. Shupyk NMA of PGE, Kyiv
  - CI of TRC Ternopil University Hospital, Lviv
  - Communal City Clinical Hospital of Ambulance, Dept of Therapy #1 D.Halytskyi Lviv NMU, Lviv
  - CI Odesa Regional Clinical Hospital, Odesa
  - SI Divisional Clinical Hospital of Uzhgorod Station of ST&BA LZ Dep of Therapy SHEI Uzhgorod NU, Uzhhorod
  - Private Small Enterprise Medical Center Pulse, Vinnytsia
  - Vinnytsya RCH for Patriotic War Invalides Therapeutic Dept # 1 Vinnytsia M.I.Pyrogov NMU, Vinnytsia
  - MCIC MC LLC Health Clinic, Vinnytsia
  - SRI of Invalid Rehabilitation (EST Complex) of Vinnytsia M.I.Pyrogov NMU MOHU, Vinnytsia
  - CI City Clinical Hospital #6 Dept of Gastroenterology, Zaporizhzhia
  - SI Branch CH of Zaporizhzhia Station-2 of SE Prydniprovska Railway Dept of Surgery Zaporizhzhia SMU, Zaporizhzhia
- United Kingdom (6):
  - Derriford Hospital, Plymouth, Devon
  - Salford Royal, Salford, Greater Manchester
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Glasgow Royal Infirmary, Glasgow, Strathclyde
  - University Hospital Coventry, Coventry, West Midlands
  - Royal Wolverhampton hospital, Wolverhampton, West Midlands

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Dulai PS, Feagan BG, Sands BE, Chen J, Lasch K, Lirio RA. Prognostic Value of Fecal Calprotectin to Inform Treat-to-Target Monitoring in Ulcerative Colitis. Clin Gastroenterol Hepatol. 2023 Feb;21(2):456-466.e7. doi: 10.1016/j.cgh.2022.07.027. Epub 2022 Aug 4. PMID 35934286
- [Derived] Peyrin-Biroulet L, Loftus EV Jr, Colombel JF, Danese S, Rogers R, Bornstein JD, Chen J, Schreiber S, Sands BE, Lirio RA. Histologic Outcomes With Vedolizumab Versus Adalimumab in Ulcerative Colitis: Results From An Efficacy and Safety Study of Vedolizumab Intravenous Compared to Adalimumab Subcutaneous in Participants With Ulcerative Colitis (VARSITY). Gastroenterology. 2021 Oct;161(4):1156-1167.e3. doi: 10.1053/j.gastro.2021.06.015. Epub 2021 Jun 16. PMID 34144047
- [Derived] Sands BE, Peyrin-Biroulet L, Loftus EV Jr, Danese S, Colombel JF, Toruner M, Jonaitis L, Abhyankar B, Chen J, Rogers R, Lirio RA, Bornstein JD, Schreiber S; VARSITY Study Group. Vedolizumab versus Adalimumab for Moderate-to-Severe Ulcerative Colitis. N Engl J Med. 2019 Sep 26;381(13):1215-1226. doi: 10.1056/NEJMoa1905725. PMID 31553834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 205 investigative sites worldwide from 29 June 2015 up to 18 January 2019.
Pre-assignment Details: Participants with a diagnosis of moderately to severely active ulcerative colitis (UC) were enrolled in a 1:1 ratio to receive vedolizumab or adalimumab and matching placebo.
Groups:
- Adalimumab SC, 160/80/40 mg: Adalimumab 160 mg, injection, subcutaneously on Day 1, adalimumab 80 mg, injection, subcutaneously at Week 2, then adalimumab 40 mg, injection, subcutaneously every 2 weeks thereafter up to Week 50. Vedolizumab placebo-matching infusion, intravenously on Day 1 and Weeks 2, 6, 14, 22, 30, 38, and 46.
- Vedolizumab IV 300 mg: Vedolizumab 300 mg, infusion, intravenously over 30 minutes on Day 1 and Weeks 2, 6, 14, 22, 30, 38, and 46. Adalimumab placebo-matching injection, subcutaneously on Day 1, Week 2, and every 2 weeks thereafter up to Week 50.
Period: Overall Study
Arm/Group | Adalimumab SC, 160/80/40 mg | Vedolizumab IV 300 mg
Started | 386 | 385
Safety Analysis Set (Participants who received at least one dose of study drug.) | 386 | 383
Completed | 217 | 270
Not Completed | 169 | 115
Not completed — Randomized but not Treated | 0 | 2
Not completed — Pretreatment Event/Adverse Event | 18 | 16
Not completed — Leukopenia or Lymphopenia | 1 | 0
Not completed — Significant Protocol Deviation | 4 | 5
Not completed — Lost to Follow-up | 14 | 4
Not completed — Voluntary Withdrawal | 39 | 41
Not completed — Pregnancy | 1 | 1
Not completed — Lack of Efficacy | 86 | 40
Not completed — Reason not Specified | 6 | 6

BASELINE CHARACTERISTICS:
Population: Randomized Set included all participants who were randomized into the study, regardless of whether they received any dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab SC, 160/80/40 mg | Vedolizumab IV 300 mg | Total
Number analyzed (Participants) | 386 | 385 | 771
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (13.44) | 40.8 (13.74) | 40.7 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 151 | 321
  Male | 216 | 234 | 450
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 39 | 23 | 62
  Unknown or Not Reported | 341 | 354 | 695
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 4 | 15
  Asian | 30 | 32 | 62
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 2 | 5
  White | 341 | 345 | 686
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 3 | 5 | 8
  Hong Kong | 1 | 4 | 5
  Korea, Republic Of | 19 | 16 | 35
  Taiwan, Province Of China | 4 | 1 | 5
  Czech Republic | 13 | 8 | 21
  Hungary | 16 | 16 | 32
  Poland | 78 | 85 | 163
  Serbia | 11 | 18 | 29
  Slovakia | 5 | 8 | 13
  Bosnia | 2 | 1 | 3
  Bulgaria | 10 | 6 | 16
  Croatia | 11 | 5 | 16
  Israel | 9 | 13 | 22
  Romania | 6 | 6 | 12
  Russia | 41 | 44 | 85
  Turkey | 9 | 5 | 14
  Ukraine | 26 | 39 | 65
  Canada | 18 | 20 | 38
  United States | 42 | 29 | 71
  Argentina | 1 | 3 | 4
  Colombia | 2 | 2 | 4
  Mexico | 9 | 3 | 12
  France | 4 | 6 | 10
  Germany | 3 | 6 | 9
  Italy | 9 | 11 | 20
  Latvia | 6 | 7 | 13
  Lithuania | 7 | 7 | 14
  Portugal | 9 | 4 | 13
  United Kingdom | 2 | 3 | 5
  Denmark | 8 | 3 | 11
  Belgium | 0 | 1 | 1
  Netherlands | 1 | 0 | 1
  Spain | 1 | 0 | 1
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed are participants with data available for height.
  cm
    number analyzed (Participants) | 386 | 383 | 769
    (all) | 170.5 (9.65) | 172.0 (9.90) | 171.3 (9.79)
Weight [Mean (Standard Deviation); unit: kg] — Population: Number analyzed are participants with data available for weight.
  kg
    number analyzed (Participants) | 386 | 383 | 769
    (all) | 73.43 (18.374) | 72.67 (16.952) | 73.05 (17.673)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is calculated from the weight taken prior to the first dose of study drug and height taken at Screening using formula, Body Mass Index = weight/[height]^2. Population: Number analyzed are participants with data available for BMI.
  kg/m^2
    number analyzed (Participants) | 386 | 383 | 769
    (all) | 25.17 (5.646) | 24.46 (4.786) | 24.82 (5.244)
Smoking Classification [Count of Participants; unit: Participants]
  Has Never Smoked | 259 | 280 | 539
  Is a Current Smoker | 23 | 19 | 42
  Is an Ex-smoker | 104 | 84 | 188
  Missing | 0 | 2 | 2
Female Reproductive Status [Count of Participants; unit: Participants] — Population: Number analyzed are female participants.
  Participants
    number analyzed (Participants) | 170 | 151 | 321
    Postmenopausal | 29 | 32 | 61
    Surgically Sterile | 18 | 17 | 35
    Female of Childbearing Potential | 123 | 102 | 225

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Clinical Remission
Description: Clinical remission was defined as a complete Mayo score of ≤2 points and no individual subscore >1 point. The Mayo score was a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consisted of 4 subscores: rectal bleeding, stool frequency, findings on endoscopy, and physician's global assessment. Each subscore was scored on a scale from 0 to 3 and the complete Mayo score ranges from 0 to 12 (higher scores indicate greater disease activity).
Time Frame: Week 52
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab SC, 160/80/40 mg | Vedolizumab IV 300 mg
Number analyzed (Participants) | 386 | 383
percentage of participants | 22.5 [18.5 to 27.0] | 31.3 [26.7 to 36.2]
Statistical Analysis 1: Comparison: Adalimumab SC, 160/80/40 mg vs Vedolizumab IV 300 mg; Test type: Superiority; p = 0.0061, Cochran-Mantel-Haenszel; Adjusted Difference = 8.8, 95% CI 2-sided [2.5 to 15.0]; P-value of the adjusted difference was based on the Cochran-Mantel-Haenszel method, stratified by concomitant use of oral corticosteroids (Yes/No) and prior use of TNF-alpha antagonist (Yes/No) or the Fisher's exact method if the numerator was <=5

2. Secondary Outcome: Percentage of Participants Who Achieved Mucosal Healing
Description: Mucosal healing was defined as a Mayo score endoscopic subscore of <= 1 point. The Mayo score was a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consisted of 4 subscores: rectal bleeding, stool frequency, findings on endoscopy, and physician's global assessment. Each subscore was scored on a scale from 0 to 3 and the complete Mayo score ranges from 0 to 12 (higher scores indicate greater disease activity).
Time Frame: Week 52
Population: FAS included all randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab SC, 160/80/40 mg | Vedolizumab IV 300 mg
Number analyzed (Participants) | 386 | 383
percentage of participants | 27.7 [23.3 to 32.5] | 39.7 [34.8 to 44.8]
Statistical Analysis 1: Comparison: Adalimumab SC, 160/80/40 mg vs Vedolizumab IV 300 mg; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel; Adjusted Difference = 11.9, 95% CI 2-sided [5.3 to 18.5]; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Who Used Oral Corticosteroids at Baseline Who Discontinued Corticosteroids and Were in Clinical Remission
Description: Corticosteroid-free remission was defined as participants using oral corticosteroids at Baseline (Week 0) who had discontinued oral corticosteroids and were in clinical remission at Week 52. Clinical remission was defined as a complete Mayo score of ≤ 2 points and no individual subscore > 1 point. The Mayo score was a standard assessment tool to measure ulcerative colitis disease activity in clinical trials. The index consisted of 4 subscores: rectal bleeding, stool frequency, findings on endoscopy, and physician's global assessment. Each subscore was scored on a scale from 0 to 3 and the complete Mayo score ranges from 0 to 12 (higher scores indicate greater disease activity).
Time Frame: Week 52
Population: Particiopants from, FAS, included all randomized participants who received at least 1 dose of study drug who used who used oral corticosteroids at Baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab SC, 160/80/40 mg | Vedolizumab IV 300 mg
Number analyzed (Participants) | 119 | 111
percentage of participants | 21.8 [14.8 to 30.4] | 12.6 [7.1 to 20.3]
Statistical Analysis 1: Comparison: Adalimumab SC, 160/80/40 mg vs Vedolizumab IV 300 mg; Test type: Superiority; p = 0.0641, Cochran-Mantel-Haenszel; Adjusted Difference = -9.3, 95% CI 2-sided [-18.9 to 0.4]; P-value of the adjusted difference was based on the Cochran-Mantel-Haenszel method, stratified by prior use of TNF-alpha antagonist (Yes/No) or the Fisher's exact method if the numerator was <=5

ADVERSE EVENTS:
Time Frame: From first dose of study drug and up to 126 days after the last dose (Up to 68 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. The safety analysis set included all participants who received at least 1 dose of study drug. Participants were analyzed according to the treatment they actually received.
Arm/Group | Adalimumab SC, 160/80/40 mg | Vedolizumab IV 300 mg
All-Cause Mortality (participants affected / at risk) | 0/386 | 1/383
Serious Adverse Events (participants affected / at risk) | 53/386 | 42/383
Other Adverse Events (participants affected / at risk) | 114/386 | 103/383
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab SC, 160/80/40 mg (N=386) | Vedolizumab IV 300 mg (N=383)
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Blindness (Eye disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 25 | 19 — One treatment-emergent death occurred during treatment with Vedolizumab IV 300 mg and was not related.
Colitis (Gastrointestinal disorders) | 1 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Therapeutic response decreased (General disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 3
Liver abscess (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Gamma-glutamyltransferase increased (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain stem haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dysgraphia (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Nerve root compression (Nervous system disorders) | 0 | 2
Major depression (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab SC, 160/80/40 mg (N=386) | Vedolizumab IV 300 mg (N=383)
Colitis ulcerative (Gastrointestinal disorders) | 42 | 26
Nasopharyngitis (Infections and infestations) | 30 | 27
Anaemia (Blood and lymphatic system disorders) | 23 | 19
Upper respiratory tract infection (Infections and infestations) | 17 | 20
Headache (Nervous system disorders) | 21 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2014-02-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT02497469/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT02497469/SAP_001.pdf